CLINICAL TRIAL: NCT05132829
Title: Azithromycin to Improve Latency in Exam Indicated Cerclage: a Randomized Control Trial
Brief Title: Azithromycin to Improve Latency in Exam Indicated Cerclage Control Trial
Acronym: ALEC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21D.746
Record Dates: First submitted 2021-10-25; First posted 2021-11-24 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Preterm Birth; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications; Physiological Effects of Drugs; Uterine Cervical Incompetence; Anti-Bacterial Agents; Azithromycin; Cefazolin
Keywords: cerclage; preterm birth; premature cervical dilation; antibiotics
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications; Uterine Cervical Incompetence | interventions — Cefazolin; Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cefazolin and Indomethacin (Other): Control arm- perioperative cefazolin and indomethacin
  Interventions: Drug: Cefazolin and indomethacin
- Azithromycin + control (Experimental): perioperative azithromycin, cefazolin and indomethacin
  Interventions: Drug: Azithromycin 1 gram IV; Drug: Cefazolin and indomethacin

INTERVENTIONS:
Drug: Azithromycin 1 gram IV — Perioperative addition of azithromycin at the time of physical exam indicated cerclage placement.
  Arms: Azithromycin + control
Drug: Cefazolin and indomethacin — Perioperative standard of care with cefazolin and indomethacin

SUMMARY:
Azithromycin is an antibiotic that is effective against bacteria that been associated with preterm birth (PTB). The purpose of this study is to evaluate if the addition of azithromycin prior to exam indicated cerclage prolongs gestation. A cerclage is a suture placed in the cervix to prolong gestation.

DETAILED DESCRIPTION:
Preterm birth (PTB) continues to be a leading cause of neonatal morbidity and mortality. The rate of spontaneous PTB (delivery before 37 weeks gestation) is one in ten pregnancies and a history of prior preterm birth remains a risk factor for recurrence. The pathophysiology of cervical insufficiency leading to PTB remains poorly understood.

While interventions for PTB prevention are limited, the American College of Obstetrics and Gynecology (ACOG) supports the use of cervical cerclage. A physical exam indicated cerclage may be placed in the setting of painless cervical dilation in the second trimester. The cerclage is believed to provide mechanical support to a weakened cervix and promote the cervical mucosal plug as a barrier to ascending infection.

While many aspects of cerclage use have been extensively studied, the use of antibiotics prior to placement remains under evaluated. While antibiotic use is recommended during cesarean section, preterm premature rupture of membranes (PPROM), and obstetric anal sphincter injuries (OASIS), ACOG currently does not recommend perioperative antibiotics or prophylactic tocolytics at the time of cerclage placement citing insufficient evidence.

Miller et al. performed a randomized controlled trial (RCT) showing an increased incidence of pregnancy prolongation by at least 28 days among women who received indomethacin and perioperative antibiotics in the setting of an exam indicated cerclage compared to those who received no perioperative medications (92.3% vs 62.5%, p=0.01). Participants in the experimental arm received cefazolin or clindamycin if they had a penicillin allergy. Cefazolin is a first generation cephalosporin that has activity against gram positive cocci and gram negative rods and is commonly used for surgical prophylaxis. Clindamycin is a protein synthesis inhibitor and covers gram positive organisms and anaerobic bacteria, making it an appropriate alternative in cases of penicillin allergy. The use of cefazolin specifically with indomethacin has been studied retrospectively and showed a significant improvement in gestational latency (adjusted relative risk [aRR] 1.21, 95% CI 1.05-1.40) and birth weight (+489.8 grams, 95% CI 64.6-915.0).

The use of prolonged azithromycin with cerclage has been studied in a prospective, non- randomized fashion. In this study, patients were given 500mg azithromycin for 3 days and this was repeated every 10 days until 34 weeks. Patients who received this regimen and a cerclage had lower PTB (65.7% vs 5.7%, p<0.001) and reduced immediate fetal mortality (37.1% vs 0%, p<0.001).

The aim of our study is to determine if the addition of azithromycin prior to exam indicated cerclage prolongs gestation. Azithromycin is a macrolide antibiotic that binds to the 50S subunit of the bacterial ribosome and inhibits transpeptidation. It is effective against a wide variety of bacteria, specifically mycoplasma which has been associated with preterm birth. Azithromycin is currently used in obstetrics for patients undergoing nonelective cesarean delivery and as part of latency antibiotics in the setting of PPROM.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton pregnancies
* ≥18 years old
* Estimated gestational age less than 24 weeks
* Meet criteria for an exam indicated cerclage
* Patients must also be able to provide consent, demonstrate an understanding of the purpose of the study, and agree to the study protocol.

Exclusion Criteria:

* Human immunodeficiency virus (HIV) positive status
* Known prolonged QT syndrome
* Major fetal congenital anomalies
* Temperature of 100.4 F or higher
* Prior cerclage during the current pregnancy
* Contraindication to indomethacin
* Allergy to both penicillin and clindamycin
* Received indomethacin or any antibiotics within 7 days before their presentation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Gestational Latency Achieved Between Cerclage Placement and Time of Delivery | 24 weeks following cerclage placement
  Mean gestational latency achieved Between Cerclage Placement and Time of Delivery

SECONDARY OUTCOMES:
Preterm birth <37 weeks, <34 weeks, <32 weeks, <28 weeks, <24 weeks | at delivery following cerclage placement. Latest will occur 26 weeks following cerclage placement.
  Preterm delivery stratified by gestational age at delivery in weeks
Mean gestational age at delivery | at delivery following cerclage placement. Latest will occur 26 weeks following cerclage placement.
  Measured in weeks
chorioamnionitis | at delivery following cerclage placement. Latest will occur 26 weeks following cerclage placement.
  Histologic or clinical diagnosis
birth weight | at delivery following cerclage placement. Latest will occur 26 weeks following cerclage placement.
  measured in grams
Admission to neonatal intensive care unit | at delivery following cerclage placement. Latest will occur 26 weeks following cerclage placement.
  If admitted, measured in days
Neonatal Morbidity and Mortality | within 28 days of delivery
  including apgars, Respiratory Distress Syndrome, Bronchopulmonary dysplasia, Retinopathy of prematurity, Intraventricular hemorrhage (IVH) (grade 3 or 4), patent ductus arteriosus, and neonatal death
Cervicovaginal cytokine analysis | Cerclage placement and 1-4 weeks after
  Measurement of proinflammatory cytokines in pg/ml (IL-1B, IL-2, IL-4, IL-6, IL-8, IL-8, IL-10, G-CSF, GM-CSF, MCP-1, TNF-a, IFN-g, CCL5, VEGF, ICAM-1) from cervicovaginal fluid at the time of cerclage placement and at follow up 1-4 weeks after placement

CONTACTS AND LOCATIONS:
Overall Officials: Jenani S Jayakumaran, MD, Principal Investigator — Thomas Jefferson University; Rupsa Boelig, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Rutgers Robert Wood Johnson, New Brunswick, New Jersey

REFERENCES:
- [Derived] Jayakumaran JS, Khanuja K, Fischer SA, Miller ES, Rosenfeld EB, Brandt JS, Piacquadio M, Kalifeh A, Boelig RC. Azithromycin to improve latency in exam-indicated cerclage: A multicenter randomized controlled trial (ALEC). Am J Obstet Gynecol MFM. 2025 Oct 22:101818. doi: 10.1016/j.ajogmf.2025.101818. Online ahead of print. PMID 41135925